CLINICAL TRIAL: NCT03257579
Title: Length of Initial Prescription at Hospital Discharge and Long-term Medication Adherence for Elderly Patients Post-Myocardial Infarction: An Interventional Study
Brief Title: Myocardial Infarction Prescription Duration Adherence Study
Acronym: MIPAD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hamilton Health Sciences Corporation (Other)
Collaborators: Population Health Research Institute (Other); Institute for Clinical Evaluative Sciences (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Health Services Research
Other Study IDs: 2979
Record Dates: First submitted 2017-06-16; First posted 2017-08-22 (Actual); Last update posted 2022-03-16 (Actual); Status verified 2022-03

CONDITIONS: Medication Adherence
Keywords: Myocardial Infarction; Adherence; Medication
MeSH Terms: conditions — Medication Adherence; Myocardial Infarction | interventions — Equipment and Supplies; Educational Status

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 90 Day Supply (Experimental): Intervention: At Hamilton Health Sciences a policy change implementing a standardized discharge prescription form of a 90-day supply with 3 repeats for all cardiac medications available on all wards where MI patients are managed.
  Interventions: Other: 90 Day Supply
- Education Alone (Experimental): At St. Joseph's Hospital and Niagara Health System education regarding the benefits of lengthening prescriptions to a 90 day supply with 3 repeats for all cardiac medications will be implemented.
  Interventions: Behavioral: Education
- Control (No Intervention): Remaining Ontario cardiac sites will receive usual care and act as concurrent control group.

INTERVENTIONS:
Other: 90 Day Supply — Policy Change implementing a 90 day standardized discharge prescription form with 3 repeats for all cardiac medications available on all wards where MI patients are managed at Hamilton Health Sciences sites
  Arms: 90 Day Supply
Behavioral: Education — Education Alone provided at St. Joseph's Hospital and Niagara Health System
  Arms: Education Alone

SUMMARY:
Quasi-experimental, controlled interrupted time series design, evaluating the impact of the intervention at Hamilton Health Sciences (HHS) where standardized prescriptions and education will be provided and St Joseph's Hospital (SJH) and Niagara Health Services (NHS) where education alone will be provided, with remaining Ontario cardiac sites as a concurrent control group.

DETAILED DESCRIPTION:
The overarching goal of this study is to reduce the morbidity and mortality of post-MI patients through improved long-term cardiac medication adherence.

The specific objectives include: 1. Assess the impact on long-term cardiac medication adherence following the implementation of a standardized increase in discharge prescription length to 90-days with 3 repeats in post-MI patients as compared to education alone and usual care; 2. Assess the cost implications of the intervention as compared to usual care; 3. Compare clinical outcomes between longer (>60 days) versus shorter prescription durations; 4. Collect baseline information to inform a multi-centre interventional study (i.e., simple monthly proportions of 1-year adherence by hospitals in Ontario).

Intervention:1. Policy Change implementing a standardized discharge prescription form available on all wards where MI patients are managed at HHS that includes a 90-day supply with 3 repeats for all cardiac medications, and education alone provided at SJH and NHS 2. Educational materials will be disseminated to all involved health care providers (e.g., physicians, residents, nurses) at the start of the intervention period to ensure the new discharge prescriptions are understood and used. Furthermore, extensive outreach to community pharmacies in LHIN IV will be undertaken with help from Ontario Pharmacists' Association (OPA) and Ontario Pharmacy Evidence Network (OPEN).

3. Education (e.g., emails, mail-outs, site visits) will recur every 3-4 months during the intervention period. Furthermore, monthly monitoring will ensure standardized prescription forms and point of care reminders are implemented at all intervention sites.

The intervention group will be exposed to this intervention post-MI and include all eligible patients at HHS/SJH/NHS in the 6-months post-intervention implementation.

ELIGIBILITY:
Inclusion Criteria:

* Use of Ontario Drug Benefits (ODB-Age >65 years, social assistance, and disability);
* Cardiac catheterization during an index admission with an MI;
* Evidence of obstructive coronary artery disease;
* Discharged alive
* Ontario Residents (Ontario, Canada)

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20896 (Actual)
Dates: Start 2017-09-05 (Actual); Primary Completion 2018-09-30 (Actual); Study Completion 2021-07-31 (Actual)

PRIMARY OUTCOMES:
Proportion of Patients with High Adherence | One year
  Increased proportion of patients with high adherence (proportion of days covered (PDC) >80%) for the combined four cardiac medications classes at one year

SECONDARY OUTCOMES:
Difference in adherence of medication classes | One year
  Difference in proportion with high adherence (mean PDC >80%) to the individual cardiac medication classes
Difference in combined and individual medications as measured by Proportion of Days Covered (PDC) | One year
  Difference in mean of Proportion of Days Covered (PDC >80%) of the combined cardiac medications as compared to PDC of individual cardiac medications classes as collected by Ontario Drug Benefits usage and reported to the Institute of Clinical Evaluative Sciences (ICES).
Discharge Prescription Length | One year
  Difference in discharge prescription length (<90 days and ≥90 days)
Clinical outcomes as measured by number of participants who experience death, myocardial infarction, coronary revascularization, and hospital readmission | One year
  Difference in proportion of participants experiencing death, myocardial infarction, coronary revascularization and hospital readmission at one year at each interventional site compared to control sites, as reported by Cardiac Care Network and analyzed by ICES.
Cost implications | One year
  Cost implications of interventions of each arm

CONTACTS AND LOCATIONS:
Overall Officials: Jon-David Schwalm, MD,FRCPC,MSc, Principal Investigator — 905-577-1423
Locations (1):
- Hamilton General Hospital, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Schwalm JD, Ivers NM, Bouck Z, Taljaard M, Natarajan MK, Nguyen F, Hijazi W, Thavorn K, Dolovich L, McCready T, O'Brien E, Grimshaw JM. Length of initial prescription at hospital discharge and long-term medication adherence for elderly, post-myocardial infarction patients: a population-based interrupted time series study. BMC Med. 2022 Jun 21;20(1):213. doi: 10.1186/s12916-022-02401-5. PMID 35725542
- [Derived] Schwalm JD, Ivers NM, Bouck Z, Taljaard M, Natarajan MK, Dolovich L, Thavorn K, McCready T, O'Brien E, Grimshaw JM. Length of Initial Prescription at Hospital Discharge and Long-Term Medication Adherence for Elderly, Post-Myocardial Infarction Patients: Protocol for an Interrupted Time Series Study. JMIR Res Protoc. 2020 Nov 4;9(11):e18981. doi: 10.2196/18981. PMID 33146624